CLINICAL TRIAL: NCT02692833
Title: Telomere Length and Telomerase Activity as a Predictor of Acute Kidney Injury Following Cardiac
Brief Title: Telomere Biology and AKI in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 010706
Record Dates: First submitted 2016-01-22; First posted 2016-02-26 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2016-09

CONDITIONS: Acute Kidney Injury; Heart Valve Diseases; Coronary Artery Disease
Keywords: Telomere; Telomerase; DNA methylation; Cell aging; Thoracic Surgery
MeSH Terms: conditions — Acute Kidney Injury; Heart Valve Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Blood samples collected for:
  Peripheral Blood Mononuclear Cells (PBMC) DNA extraction from buffy coat Right atrial tissue samples (subset) Urine and plasma/serum for urinary biomarkers (subset)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AKI Patients: Patients who develop acute kidney injury within the first 5 days following their cardiac surgical operation.
  Interventions: Other: No intervention
- Non-AKI patients: Patients who do not develop acute kidney injury within the first 5 days following their cardiac surgical operation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. This is an observational study of how patients' renal function responds to their surgery. The groups are defined by this response. There is no difference between clinical interventions between the two groups.

SUMMARY:
The purpose of this study is to investigate whether biomarkers of cell senescence and aging can predict the development of acute kidney injury following cardiac surgery.

DETAILED DESCRIPTION:
Patients with pre-operative renal dysfunction are at increased risk of developing cardiac surgery associated acute kidney injury (AKI) but a proportion of patients with normal kidney function will also be affected. Studies show that patients developing AKI post cardiac surgery have a poorer long term prognosis, even if their kidney function subsequently returns to normal However, the cause for this is not currently understood. We postulate that a unifying mechanism makes such patients more susceptible to developing post-operative AKI and of having an overall worse long term prognosis. We suggest that this mechanism is reduced regenerative capacity of tissues. To test this hypothesis we will measure several markers of cell senescence and aging including telomere length, telomerase activity, and DNA methylation status.

Previous animal studies have shown that reduced telomere length and telomerase activity in mice increases their susceptibility to ischaemia induced renal injury. The current study will look at whether a similar association is seen in humans, using cardiopulmonary bypass as a mechanism for studying ischaemia/inflammatory induced kidney injury. It aims to answer the primary research question: Are telomere length and telomerase activity related to the development of acute kidney injury following cardiac surgery? The presence of such an association would provide new avenues in the development of biomarkers to predict outcomes following cardiac surgery. In addition to scoring tools currently in clinical practice, such biomarkers might allow better risk stratification of patients undergoing cardiac surgery.

Patient Registry and sample storage: Tissue samples and patient data collected in these patients will also form part of the Barts Cardiovascular Registry (BAR). This is a Biobank facility run by Barts Heart Centre in collaboration with United Kingdom (UK) Biobank. All aspects of patient recruitment, data collection, data storage, and data analysis will be covered by Standard Operating Procedures to ensure data quality of the registry.

Quality assurance: The management team for the BAR will be responsible for auditing the completeness and validity of the data.

Sample size: As we have no preceding data on a possible association with telomere biology and AKI post-cardiac surgery we have been unable to perform a power calculation for sample size. In effect, the present study will be a large pilot study looking at this association. Previously reported studies give an incidence of AKI following cardiac surgery of between 15 and 25%. In order to have approximately 200 AKI patients to study, we will aim to recruit 1000 patients. This is realistic given that the Barts Heart Centre should be performing approximately 50 cardiac operations per week. Once recruitment is established, an interim analysis will be performed to allow a more accurate estimation of sample size.

Statistical analysis: All relevant clinical parameters will be analysed by frequencies, tabulations, correlations, distributions of normality and comparisons accordingly. An array of statistical methods will be employed for parametric and non-parametric data including Multivariate of all factors associated with the development of acute kidney injury following cardiac surgery. Receiver operator characteristic (ROC) curve analysis will be used to investigate clinical outcomes and the new markers of cell senescence (telomere length, telomerase activity, and DNA methylation status). Missing data values will be rectified where possible by review of the primary medical records. Missing data values due to incomplete sample collection will be dealt with by statistical modelling.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing cardiac surgery at Barts Heart Centre

Exclusion Criteria:

* Renal dialysis patients
* Renal transplant patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 5 days
  The development of acute kidney injury in the first 5 days of surgery.

SECONDARY OUTCOMES:
In hospital mortality | 30 days
  All cause death during the post-operative hospital stay or within 30 days whichever is sooner.
Major adverse cardiac and cerebrovascular events | 30 days
  Covers several outcomes within the index hospital admission of within 30 days whichever is shorter. The included outcomes are: Cardiac related mortality, stroke, myocardial infarction, and need for repeat revascularisation.
length of stay | Will be assessed upon patient's discharge from hospital. Typically 5-10 days but variable
  length of in-hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Magdi M Yaqoob, PhD, Study Director — Queen mary Univerisity of London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data outside of our research group

REFERENCES:
- [Background] Thakar CV, Arrigain S, Worley S, Yared JP, Paganini EP. A clinical score to predict acute renal failure after cardiac surgery. J Am Soc Nephrol. 2005 Jan;16(1):162-8. doi: 10.1681/ASN.2004040331. Epub 2004 Nov 24. PMID 15563569
- [Background] Hobson CE, Yavas S, Segal MS, Schold JD, Tribble CG, Layon AJ, Bihorac A. Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery. Circulation. 2009 May 12;119(18):2444-53. doi: 10.1161/CIRCULATIONAHA.108.800011. Epub 2009 Apr 27. PMID 19398670
- [Background] Loef BG, Epema AH, Smilde TD, Henning RH, Ebels T, Navis G, Stegeman CA. Immediate postoperative renal function deterioration in cardiac surgical patients predicts in-hospital mortality and long-term survival. J Am Soc Nephrol. 2005 Jan;16(1):195-200. doi: 10.1681/ASN.2003100875. Epub 2004 Nov 24. PMID 15563558
- [Background] Westhoff JH, Schildhorn C, Jacobi C, Homme M, Hartner A, Braun H, Kryzer C, Wang C, von Zglinicki T, Kranzlin B, Gretz N, Melk A. Telomere shortening reduces regenerative capacity after acute kidney injury. J Am Soc Nephrol. 2010 Feb;21(2):327-36. doi: 10.1681/ASN.2009010072. Epub 2009 Dec 3. PMID 19959722